CLINICAL TRIAL: NCT01031979
Title: Psychophysiology of Prolonged Exposure for PTSD With/Without Yohimbine
Brief Title: Prolonged Exposure for Post Traumatic Stress Disorder (PTSD) With/Without Yohimbine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDA-2-013-09F
Record Dates: First submitted 2009-12-04; First posted 2009-12-15 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; Prolonged Exposure; extinction; habituation; psychophysiology
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders | interventions — Yohimbine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Yohimbime Group (Experimental): Patients will take one 21.6 mg. dose of yohimbine one hour before first imaginal exposure in PE.
  Interventions: Drug: Yohimbine
- Placebo Group (Placebo Comparator): Patients will take a placebo one hour before first imaginal exposure in PE.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Yohimbine — alpha-2 adrenergic receptor antagonist
  Arms: Yohimbime Group
Drug: Placebo — Placebo
  Arms: Placebo Group

SUMMARY:
The proposed study has three distinct but related research objectives. The first goal is to measure physiological correlates of successful treatment with Prolonged Exposure (PE) therapy for posttraumatic stress disorder (PTSD) in veterans of the Iraq and Afghanistan wars. Individuals with PTSD often experience elevated heart rates and other objectively measurable signs of anxiety when confronted with safe situations that remind them of past dangerous situations. We will measure physiological responses and compare the outcomes to patient's self reported subjective accounts of symptom improvement on traditional measures of PTSD. Developing a way to measure objective gains in symptoms improvement may help researchers who are studying ways to improve PTSD treatment. The second goal of the study is to investigate if yohimbine, a drug found to promote a specific type of learning, will improve treatment outcomes for veterans in PTSD treatment. The third goal is to investigate if ability to get used to loud startling audio tones correlates to baseline PTSD pathology and treatment outcomes for PE. This goal represents an important step forward in understanding characteristics of heritable traits that are related PTSD. It is significant because such research may one day lead to the development of individual responder policies that will assist patients by individualizing treatment plans based on personal characteristics.

DETAILED DESCRIPTION:
The proposed study has three distinct but related research objectives. The first research goal is to measure psychophysiological correlates of treatment gains associated with Prolonged Exposure (PE) therapy for PTSD in veterans of Operations Enduring Freedom and Iraqi Freedom (OEF/OIF). Specifically, heart rate, heart rate variability, skin conductance, and facial electromyography, will be recorded before and after treatment during a three minute anxiety probe specific to the patient's index trauma. These measures will be compared to patient's self reported subjective accounts of symptom improvement on traditional measures of PTSD pathology (Subjective Units of Distress (SUDs), PTSD Checklist-Military Version (PCL), Clinician Administered PTSD Scale (CAPS), and the Beck Depression Inventory (BDI)). This goal is significant for veterans because currently no widely used objective criteria exist to measure treatment progress in PTSD. While the preponderance of existing evidence suggests that no one objective psychophysiological measurement will be a valid correlate for all individuals, even establishing a measurement paradigm that can show mean differences between groups will provide researchers with an objective tool to measure outcomes on clinical trials.

The second goal of the study is to investigate if the administration of yohimbine, a drug found to promote the extinction of conditioned fear in animal models, and more recently, in humans with claustrophobia, improves the facilitation of fear extinction in PE. Yohimbine is a safe drug that is already extensively used in human populations. Specifically, this goal will be investigated using a double blind placebo controlled randomized trial design. The hypothesis is that one 21mg oral dose of yohimbine given concurrently with a 40 minute imaginal exposure exercise in PE will lead to a greater reduction in cue-induced anxiety during the following weekly PE session than placebo. This goal is significant because current projections of PTSD in OEF/OIF veterans indicate that the need for psychological services will likely outpace the supply of such services. Accordingly, assisting treatments to be more efficient will likely translate into more veterans receiving much needed mental health services.

The 3rd goal is to investigate if ability to habituate to loud, 95db, audio tones correlates to baseline PTSD pathology and treatment outcomes for PE. This goal represents an important step forward in understanding characteristics of trait habituation, fear extinction, and learning in humans, which are all factors related to the successful treatment of PTSD. It is also significant because such research may lead to the development of individual responder policies that will assist veterans by individualizing treatment plans based on personal characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be competent to provide informed consent for research participation.
* Subjects must be male veterans and post deployed active duty male personnel of OEF/OIF.
* Subjects must be between the ages of 18 and 45.
* Subjects must meet DSM-IV diagnostic criteria for PTSD on the CAPS.
* For subjects taking SSRI's, subjects must be stabilized on the current prescribed dose for a period of at least 14 days prior to the trial and remain at that dose for the remainder of the study. Subjects who change their SSRI status or dosage during the study will continue to receive services via the study resources but data generated will not be used in analyses. Subjects will be eligible for the study if they are willing to titrate off potentially confounding agents prior to yohimbine administration (for a period of five half-lives), given that such titration is also clinically appropriate and deemed to be in the patient's best interests.

Exclusion Criteria:

* Subjects with a recent (< 2 month) history of psychiatric hospitalization or suicide attempt. Recent work with veterans with severe mental illness suggests that a 2-month period of stabilization is sufficient to minimize risk and possible relapse (Frueh, 2005). Subjects with an existing diagnosis of schizophrenia or other Axis I serious mental illnesses (SMI, besides PTSD) will be excluded. SMI will include any severe and persistent mental illness.
* Subjects with a current diagnosis of drug dependence, due to potential interactions with study measurements and treatments. Alcohol use disorders will be allowed given that subjects can pass exclusion criterion 12 without withdrawal symptoms.
* Subjects with any acute illness or fever. Individuals who otherwise meet study criteria will be rescheduled for evaluation for participation.
* Subjects with evidence of or a history of clinically significant hematological, endocrine, cardiovascular, hepatic, pulmonary, renal, gastrointestinal, or neurological disease including diabetes, as these conditions may affect physiological/subjective responses.
* Subjects with SCID-diagnosed panic disorder, as yohimbine may precipitate panic attacks.
* Subjects with an abnormal ECG.
* Subjects with a blood pressure of 140/90 or higher, as yohimbine has been shown to elevate blood pressure.
* Subjects taking Beta blockers, alpha-adrenergic agents, Beta-agonist inhalers, opiates or opiate antagonists and any psychotropic medications other than SSRI's because these may affect test response.
* Subjects who are unwilling or unable to maintain abstinence for three days prior to yohimbine administration from over-the-counter drugs with sympathomimetic properties, e.g., asthma medications, cold medicines with ephedrine, dietary supplements with ephedrine alkaloids, and illegal drugs, e.g., amphetamines, methamphetamine, cocaine, and MNDA as well as alcohol because these may exacerbate the action of yohimbine.
* Subjects taking alpha-adrenergic antagonists, e.g. prazosin for hypertension; and beta-adrenergic antagonists, e.g. propranolol. Because they may attenuate effects of yohimbine. Subjects will be eligible for the study if they are willing to titrate off potentially confounding agents prior to yohimbine administration (for a period of five half-lives), given that such titration is also clinically appropriate and deemed to be in the patient's best interests.
* Asthmatic subjects and subjects on medications for hypertension, due to criteria 9 and 10.

These inclusion/exclusion criteria will allow the majority of veterans treated in the PCT to be study eligible. Accordingly, the sample will be likely generalizable to the population of interest.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Males only.
Enrollment: 26 (Actual)
Dates: Start 2010-12-01 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2015-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter W. Tuerk, PhD MA BA, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keller SM, Tuerk PW. Evidence-based psychotherapy (EBP) non-initiation among veterans offered an EBP for posttraumatic stress disorder. Psychol Serv. 2016 Feb;13(1):42-8. doi: 10.1037/ser0000064. Epub 2015 Dec 14. PMID 26654474
- [Derived] Yuen EK, Gros DF, Price M, Zeigler S, Tuerk PW, Foa EB, Acierno R. Randomized Controlled Trial of Home-Based Telehealth Versus In-Person Prolonged Exposure for Combat-Related PTSD in Veterans: Preliminary Results. J Clin Psychol. 2015 Jun;71(6):500-12. doi: 10.1002/jclp.22168. Epub 2015 Mar 25. PMID 25809565

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Yohimbime Group | Placebo Group
Started | 14 (To meet eligibility requirements for randomization, subjects had to reach session 3 w/o dropping.) | 12 (To meet eligibility requirements for randomization, subjects had to reach session 3 w/o dropping.)
Completed Primary Outcome Measure | 12 | 12
Completed | 9 (These are individuals who completed treatment in the study.) | 8 (These are individuals who completed treatment in the study.)
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 5 | 4

BASELINE CHARACTERISTICS:
Population: 14 participants were randomized to the yohimbine group; however only 12 completed the primary outcome assessment at session 4 and were able to be analyzed.
Groups:
- Yohimbine Group: Patients will take one 21.6 mg. dose of yohimbine one hour before first imaginal exposure in PE.
  Yohimbine: alpha-2 adrenergic receptor antagonist
- Total: Total of all reporting groups
Arm/Group | Yohimbine Group | Placebo Group | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 34.6 [18 to 45] | 29.9 [18 to 45] | 32.4 [18 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Trauma-Cued Heart Rate Reactivity
Description: The primary outcome was trauma-cued heart rate reactivity a week after the drug visit as measured by the PTSD Brief Reactivity (PBR) task. For each patient, a 3-minute trauma script was constructed containing vivid details of the target trauma and used in tandem with a standard neutral script for baseline measurement. Heart rate reactivity for each time point was the beats per minute (BPM) difference between the neutral and trauma scripts represented as a slope.
Time Frame: One week after drug visit
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Yohimbine Group | Placebo Group
Number analyzed (Participants) | 14 | 12
beats per minute | 71.01 (3.84) | 75.08 (3.11)
Statistical Analysis 1: Comparison: Yohimbine Group vs Placebo Group; Test type: Superiority or Other; p < 0.001, mixed effects/hierarchical linear model; Beta = -1.44, 95% CI 2-sided [-2.29 to -0.59]

2. Secondary Outcome: Change in Clinician Administered PTSD Scale (CAPS) Score
Description: The CAPS is a structured interview for diagnosis of PTSD and is widely considered the gold-standard assessment. The CAPS produces a total score ranging from 0-136, with higher scores indicating more severe PTSD symptom severity. A 15-point decrease is considered clinically significant.
Time Frame: 0 Weeks, 15 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yohimbine Group | Placebo Group
Number analyzed (Participants) | 12 | 12
units on a scale
  Baseline CAPS | 67.33 (24.49) | 65.00 (13.01)
  Week 15 CAPS (post-treatment) | 25.13 (14.93) | 20.62 (10.84)
Statistical Analysis 1: Comparison: Yohimbine Group vs Placebo Group; Test type: Superiority or Other; p = .39, Hierarchical Linear Modeling; Slope = -0.87

3. Secondary Outcome: Change in Post Traumatic Stress Disorder Checklist (PCL) Score
Description: The PCL is a 17-item self-report measure of PTSD symptom severity based on the DSM-IV and has adequate psychometric properties. The PCL produces a score range between 17-85, with higher scores indicating more distress related to PTSD symptoms. A 10-point decrease on the PCL is considered clinically significant.
Time Frame: 0 weeks, 15 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yohimbine Group | Placebo Group
Number analyzed (Participants) | 12 | 12
units on a scale
  Baseline PCL | 64.00 (12.49) | 60.25 (14.53)
  Week 15 PCL (post-treatment) | 27.37 (6.63) | 28.50 (8.88)
Statistical Analysis 1: Comparison: Yohimbine Group vs Placebo Group; Test type: Superiority or Other; p = .58, Hierarchical Linear Modeling; Slope = -0.55

4. Secondary Outcome: Change in Becks Depression Inventory (BDI-II) Score
Description: The BDI-II is a 21-item self-report measure that assesses depressive behavioral symptoms. It has demonstrated adequate psychometric validity, and external validity and is used widely as the dependent variable in treatment outcomes research. The BDI-II produces score ranges from 0-63, with higher scores indicating more severe depression symptom severity. A 5-point decrease on the BDI-II is considered clinically significant.
Time Frame: 0 weeks, 15 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yohimbine Group | Placebo Group
Number analyzed (Participants) | 12 | 12
units on a scale
  Baseline BDI-II | 30.56 (13.10) | 22.62 (7.05)
  Week 15 BDI-II (post-treatment) | 7.00 (5.68) | 7.87 (7.97)
Statistical Analysis 1: Comparison: Yohimbine Group vs Placebo Group; Test type: Superiority or Other; p = .03, Hierarchical Linear Modeling; Beta = -1.60, 95% CI 2-sided [-2.71 to -0.49]

ADVERSE EVENTS:
Arm/Group | Yohimbine Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes